CLINICAL TRIAL: NCT04547439
Title: Sleep and Circadian Regulation in Diabetic Retinopathy: The Role of Intrinsically Photosensitive Retinal Ganglion Cells and Melatonin Supplementation
Brief Title: Sleep, Diabetic Retinopathy and Melatonin
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: University of Chicago (Other)
Responsible Party: Principal Investigator, Sirimon Reutrakul, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2020-1052
Record Dates: First submitted 2020-06-27; First posted 2020-09-14 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Double blinded randomized controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and investigators are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Active Comparator): Placebo
  Interventions: Other: Placebo
- Melatonin (Active Comparator): Melatonin
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — Melatonin 3 mg will be taken nightly for 8 weeks
  Arms: Melatonin
Other: Placebo — Placebo will be given nightly for 8 weeks
  Arms: Control

SUMMARY:
This study explores the use of melatonin in patients with diabetic retinopathy

DETAILED DESCRIPTION:
This is a randomized controlled study using melatonin for 8 weeks in patients with diabetic retinopathy on outcomes of sleep and circadian regulation

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (clinically diagnosed, taking anti-diabetes medications or history of elevated A1C≥6.5%)
* 40-65 years of age
* Diabetic retinopathy of at least moderate degree

Exclusion Criteria:

* use of melatonin
* antidepressants or antipsychotics
* illicit drug use
* night shift work or travel beyond 2 time zones in the month before enrollment
* end stage renal disease requiring renal replacement therapy
* history of stroke or transient ischemic attacks
* history of dementia or memory impairment
* uncontrolled congestive heart failure or recent hospitalization for cardiac condition (6 months)
* chronic obstructive pulmonary disease requiring oxygen
* severe chronic liver disease such as cirrhosis
* ongoing treatment for major medical problems such as cancer
* history of severe hypoglycemia defined as hypoglycemic episodes requiring assistance from others within the past six months.
* Significant depressive symptoms
* untreated severe OSA (AHI≥ 30 events/hour),
* uncontrolled hypertension (blood pressure ≥ 160/100 mmHg),
* uncontrolled diabetes (A1C ≥ 11%),
* abnormal TSH
* abnormal liver function (AST or ALT>3x upper limits of normal
* use of sedatives and hypnotics.
* clinically significant epiretinal membranes, clinically significant lens opacities, or cystoid macular edema, iris neovascularization, iris atrophy, or an asymmetrically shaped pupil, nuclear sclerotic, posterior subcapsular, or cortical lens opacities greater than 2+, a history of pan-retinal photocoagulation.
* hemoglobin <11.5 g/dL in women and <13.5 g/dL in men.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Sleep pattern | 14 days
  Sleep pattern: Sleep duration and sleep efficiency will be assessed by wrist actigraphy, to be worn by the participants for 14 days
Melatonin and Cortisol Rhythm | 24 hours
  Melatonin and cortisol pattern (peak times of the levels, dim light melatonin onset) will be assessed from 24 hour blood sampling

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brzezinski A, Vangel MG, Wurtman RJ, Norrie G, Zhdanova I, Ben-Shushan A, Ford I. Effects of exogenous melatonin on sleep: a meta-analysis. Sleep Med Rev. 2005 Feb;9(1):41-50. doi: 10.1016/j.smrv.2004.06.004. PMID 15649737
- [Background] Singer C, Tractenberg RE, Kaye J, Schafer K, Gamst A, Grundman M, Thomas R, Thal LJ; Alzheimer's Disease Cooperative Study. A multicenter, placebo-controlled trial of melatonin for sleep disturbance in Alzheimer's disease. Sleep. 2003 Nov 1;26(7):893-901. doi: 10.1093/sleep/26.7.893. PMID 14655926
- [Background] Garfinkel D, Laudon M, Nof D, Zisapel N. Improvement of sleep quality in elderly people by controlled-release melatonin. Lancet. 1995 Aug 26;346(8974):541-4. doi: 10.1016/s0140-6736(95)91382-3. PMID 7658780
- [Background] Raygan F, Ostadmohammadi V, Bahmani F, Reiter RJ, Asemi Z. Melatonin administration lowers biomarkers of oxidative stress and cardio-metabolic risk in type 2 diabetic patients with coronary heart disease: A randomized, double-blind, placebo-controlled trial. Clin Nutr. 2019 Feb;38(1):191-196. doi: 10.1016/j.clnu.2017.12.004. Epub 2017 Dec 12. PMID 29275919